CLINICAL TRIAL: NCT03302052
Title: Investigation About Advance Directives
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DRAPE
Record Dates: First submitted 2017-10-01; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Advance Directive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Advance directives are again in the heart of debate since the Leonetti-Claeys's law . These pieces of legislation allow everyone to decide by advance their wishes of the end of life.However, it does not seem that to legislate on a subject is enough to apply the text of law. High authority of health suggest that medical and paramedical staff have to participate to the elaboration of the questionnaire and the redaction of advance directives.

So the aim is that ,before asking patient about their knowledge on these advance directive, to evaluate if the staff knows about the law .

ELIGIBILITY:
Inclusion Criteria:

* nurse
* doctors
* paramedical staff

Exclusion Criteria:

* refusing participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Every medical and paramedical staff of St JOSEPH'S Hospital (Paris)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Scoring the degree of knowledge of the staffs and doctors of the GHPSJ | 1 day
  every staff and doctors have to answer to a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France